CLINICAL TRIAL: NCT07263230
Title: An Open-label Single Center Study Evaluating the Safety and Efficacy of Roflumilast Foam 0.3% in Subjects With Hidradenitis Suppurativa
Brief Title: The Safety and Efficacy of Roflumilast Foam in HS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Martina Porter, Vice Chair of Dermatology Research, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000987
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: HS; Hidradenitis Suppurativa; Roflumilast; Topical medication
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Roflumilast 0.3% topical foam (Experimental): Roflumilast 0.3% topical foam to be applied QD to all active fields for the duration of the 16-week trial.
  Interventions: Drug: Roflumilast 0.3% topical foam

INTERVENTIONS:
Drug: Roflumilast 0.3% topical foam — Roflumilast foam, 0.3%, is a phosphodiesterase 4 inhibitor
  Other Names: ZORYVE

SUMMARY:
This study investigates the efficacy of topical roflumilast foam in patients with HS.

DETAILED DESCRIPTION:
Hidradenitis Suppurativa (HS) is a chronic inflammatory skin condition that causes painful and inflamed lumps and abscesses often in the underarms, groin and buttocks. The purpose of this study is to assess the safety and efficacy of QD 0.3% topical roflumilast foam in patients with HS over 16 weeks, with or without previous treatment. The drug involved in this study, 0.3% topical roflumilast foam, is investigational.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older
2. Participants are legally competent to sign and give informed consent.
3. Diagnosis of HS based on clinical history and physical examination for at least 3 months.
4. Diagnosis of HS (Hurley I or II) with a total AN count of at least 4 to ≤ 10, with no draining tunnels at screening and baseline visits with an AN of >4 affecting at least one distinct anatomical region.
5. Agreement to NOT use topical and systemic antibiotics and intralesional steroids for treatment of HS during the study.
6. Agreement to NOT use a diluted beach bath or topical antiseptic washes containing chlorhexidine gluconate or benzoyl peroxide on the areas affected by HS lesions during the study.
7. Subjects who have had surgery in the treatment area should be at least 3 months post procedure (this applies to deroofing/ marsupialization or excision, not incision & drainage)
8. Females of childbearing potential (FOCBP) must have a negative urine pregnancy test at Screening and Baseline/Day 1. In addition, sexually active FOCBP must agree to use at least one form of a highly effective or barrier method of contraception throughout the trial. The use of abstinence as a contraceptive measure is acceptable if this is a consistent part of a lifestyle choice and an acceptable backup method has been identified if the subject becomes sexually active.
9. Females of non-childbearing potential should be post-menopausal with spontaneous amenorrhea for at least 12 months or have undergone surgical sterilization (permanent sterilization methods include hysterectomy, bilateral oophorectomy, hysteroscopic sterilization, bilateral tubal ligation or bilateral salpingectomy).
10. In good health as judged by the Investigator, based on medical history, targeted physical examination, and vital signs. Subjects and parent(s)/legal guardian(s) are considered reliable and capable of adhering to the Protocol and visit schedule, according to the judgment of the Investigator.

Exclusion Criteria:

1. Subjects with any medical condition or physical examination abnormality that would prevent study participation or place the subject at significant risk, as judged by the Investigator
2. Subjects who cannot discontinue medications and treatments prior to the Baseline visit and during the study according to Excluded Medications and Treatments (see table of Excluded Medications and Treatments with washout timelines).
3. Presence of draining tunnels at screening or at baseline visits
4. Subjects who are unwilling to refrain from prolonged sun exposure and from using a tanning bed or other artificial light emitting devices (LEDs) for 4 weeks prior to Baseline/Day 1 and during the study.
5. Subjects with skin conditions other than HS that would interfere with evaluations of the effect of the study medication on HS, as determined by the Investigator.
6. Subjects with any condition on the treatment area which, in the opinion of the Investigator, could confound efficacy measurements.
7. Known allergies to excipients in Roflumilast foam (petrolatum, isopropyl palmitate, methylparaben, propylparaben, diethylene glycol monoethyl ether, hexylene glycol, cetylstearyl alcohol, dicetyl phosphase and ceteth-10 phosphate).
8. Subjects who cannot discontinue the use of systemic CYP3A4 inhibitors or dual inhibitors that inhibit both CYP3A4 and CYP1A2 simultaneously for 2 weeks prior to Baseline/Day 1 and during the study period.
9. Subjects who have received oral roflumilast (Daxas®, Daliresp®) within 4 weeks prior to Baseline/ Day 1.
10. History of severe depression, suicidal ideation or behavior at Baseline/Screening
11. Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
12. Previous treatment with Roflumilast cream or foam (any potency) or current Roflumilast use for any other indication at the baseline visit that would be expected to continue during the trial.
13. Subjects with a history of major surgery within 4 weeks prior to Baseline/Day 1 or subjects who have major surgery planned during the study.
14. Subjects with a history of chronic alcohol or drug abuse within 6 months prior to Screening.
15. Current or a history of cancer within 5 years except for fully treated skin basal cell carcinoma, cutaneous squamous cell carcinoma or carcinoma in situ of the cervix.
16. Parent(s)/legal guardian(s) who are unable to communicate, read, or understand the local language(s). Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.
17. Subjects who are family members of the clinical study site, clinical study staff, or sponsor, or family members of enrolled subjects living in the same house.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Abscess and Inflammatory Nodule (AN) Count at Week 16. | Baseline and Week 16
  Change from Baseline was calculated as the Week 16 value minus the Baseline value. Baseline counts were defined as abscesses and/or inflammatory nodules present at Baseline, any new nodules identified after baseline were not counted.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Porter, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No